CLINICAL TRIAL: NCT02424448
Title: BIOMETHS Study. A Methodology Study to Determine the Feasibility, Evaluability and Temporal Variability in Candidate Pharmacodynamic Markers of Drug Action in Castration Resistant Prostate Cancer
Brief Title: Study to Determine the Feasibility, Evaluability and Variability in Markers of Drug Action in Castration Resistant Prostate Cancer
Acronym: BIOMETHS
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Safia Barber, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Other Study IDs: CFTSp063 / 12_DOG04_145
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Original diagnostic tumour blocks will be returned at the end of the study. Biopsy samples taken will either be retained or disposed of when the study is completed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Metastatic CRPC: Patients with metastatic prostate cancer post maximal androgen blockade (MAB) with primary or metastatic cancer deposits amenable to biopsy. Patients will have biopsies, blood and urine samples taken.
  Interventions: Procedure: Biopsies, blood and urine samples

INTERVENTIONS:
Procedure: Biopsies, blood and urine samples — Session 1: Biopsies will be taken from the main study lesion and up to 2 metastatic sites at 1 visit or over 3 visits. Both formalin fixed and snap frozen material will be collected. At the session (i.e. once over the potential maximum of 3 visits in a session) a urine sample, blood samples for circulating tumour cells (CTC) and an exploratory blood sample (processed to plasma) will be taken.
  Session 2: 7 days +/-3 following the last biopsy taken from Session 1, repeat biopsies from the same tumour sites will be obtained. In cases where this is not possible, it is acceptable to biopsy alternative lesions. As in Session 1 biopsies may be taken at 1 visit or over 3 visits and urine, CTC blood samples and an exploratory blood sample (processed to plasma) will be taken.

SUMMARY:
This is a biopsy feasibility study in which patients with castration resistant prostate cancer (CRPC) will be asked to donate primary and metastatic tumour tissue (both archival and de novo), blood samples, a urine specimen and clinical data for research.

DETAILED DESCRIPTION:
The study aims to determine the feasibility of sampling and evaluability of biomarkers in CRPC tissue samples and circulating tumour cells (CTCs). Exploratory biomarker analysis may include, but will not be limited to, understanding the potential proof of mechanism (POM), proof of principle (POP) or predictive biomarkers of response to potential therapeutic agents for CRPC patients, or factors that may influence the development of CRPC.

This study is predicated on the continued development of agents targeting the PI3K pathway such as AZD(AstraZeneca Drug)8186 (PI3Kb); AZD5363 (Akt) and AZD2014 (mTOR) and anti-hormonals which are expected to deliver benefit in the management of tumours dependent on PI3K signalling as a result of e.g. phosphatase and tensin homolog (PTEN) deficiency or androgen receptor activation.

Loss of PTEN is common in CRPC. Current data indicate that AZD8186 inhibits PI3K downstream signalling in PTEN deficient but not in PTEN proficient cells and hence POM and efficacy will need to be determined in tumours with PTEN protein loss. In future studies, paired biopsy tumour tissue will be accessible for assessment of POM and PTEN status, either bone metastases lymph node metastases, or within the prostate tumour.

Recruitment of patients will be carried out in two stages as follows:

Stage 1 The first 10 eligible and consenting patients will be enrolled in the study and will undergo sequential biopsies. For all stage one participants, the PTEN status will be retrospectively determined from archival tumour samples by immuno-histochemistry (IHC).

The results of the PTEN analysis from Stage 1, will determine the number of patients in Stage 2 that must be PTEN positive or PTEN null. For this study the intent is to have equal numbers of each type i.e. ten PTEN positive and ten PTEN null.

Stage 2

In Stage 2, patients will be asked to sign a pre-screening consent form for their archival tumour sample to be analysed for PTEN status prior to undergoing any main study screening procedures. If their PTEN status matches one of the available slots they will be enrolled into the study.

Once a cohort reaches ten PTEN positive and ten PTEN null patients, it will close to recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic prostate cancer post maximal androgen blockade (MAB) with primary or metastatic cancer deposits amenable to biopsy
* Patients aged 18 years and older
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* World Health Organisation (WHO) performance status 0 to 2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
* Provision of archival tumour sample for PTEN status determination as directs group assignment
* Provision of written informed consent
* Provision of cancer tissue samples, willing to undergo 1-3 biopsies on 2 separate occasions
* No change of cancer treatment anticipated until final biopsy/ blood samples have been taken
* Serum testosterone level <50 ng/dL sustained by medical or surgical castration

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrolment in the present study
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that made it undesirable for the patient to participate in the study
* Any investigational agents or study drugs from a previous clinical study within 30 days of the first tissue collection
* Radiotherapy to lesion to be biopsied within 4 weeks of biopsy
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Patients at increased risk of bleeding as a result of biopsy
* History of bleeding disorders or thrombocytopenia (platelets <100)
* Concomitant treatment with anticoagulant therapy such as warfarin/low molecular weight heparin (Aspirin not contra-indicated but consider temporary cessation if biopsy site has higher risk of bleeding e.g. liver)
* Current urinary tract infection (UTI) or prostatitis
* Known infection with HIV, Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males (18+) with metastatic hormone refractory prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of formalin fixed cancer tissue samples evaluable for immunohistochemical analysis | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
Baseline levels of biomarkers in formalin fixed cancer tissue samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
Intra-lesion temporal variability between formalin fixed cancer tissue samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
Intra-lesion spatial variability between formalin fixed cancer tissue samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)

SECONDARY OUTCOMES:
Percentage of frozen cancer tissue samples evaluable for biomarker analysis | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
Baseline levels of biomarkers in frozen cancer tissue samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
Intra-lesion temporal variability between frozen cancer tissue samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
Intra-lesion spatial variability between frozen cancer tissue samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)

OTHER OUTCOMES:
Intra-patient, inter-lesion variability (where possible) between samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
Percentage concordance between biomarker measurements on circulating tumour cells (CTCs) and tumour samples | Samples taken in session 1 (1 to 3 visits) and then 7 days +/- 3 days at session 2 (1 to 3 visits)
  (1 to 3 visits)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Elliott, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom